CLINICAL TRIAL: NCT02524171
Title: Improving Treatment Engagement and Outcomes Among Justice-involved Veterans
Brief Title: Justice-Involved Veterans and Moral Reconation Therapy
Acronym: MRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 14-081
Record Dates: First submitted 2015-08-05; First posted 2015-08-14 (Estimated); Results first posted 2021-12-20 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Antisocial Personality Disorder; Substance Use Disorder
Keywords: crime; mental health; substance abuse; homelessness; Veterans
MeSH Terms: conditions — Antisocial Personality Disorder; Substance-Related Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research Assistants conducting the 6- and 12- month outcome assessments are blinded to condition assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moral Reconation Therapy (MRT) (Experimental): MRT is a group-based cognitive-behavioral intervention to restructure antisocial thinking. Patients will receive two groups per week of this intervention for approximately 12 weeks, in addition to the usual care they receive in the mental health residential rehabilitation treatment program.
  Interventions: Behavioral: Moral Reconation Therapy (MRT)
- Usual Care (UC) (No Intervention): Usual care provided by the mental health residential rehabilitation treatment programs, which patients in both groups are in.

INTERVENTIONS:
Behavioral: Moral Reconation Therapy (MRT) — MRT is a group-based cognitive-behavioral intervention to restructure antisocial thinking. Patients will receive two groups per week of this intervention for approximately 12 weeks, in addition to the usual care they receive in the mental health residential rehabilitation treatment program.
  Other Names: MRT
  Arms: Moral Reconation Therapy (MRT)

SUMMARY:
The purpose of this study is to determine whether Moral Reconation Therapy (MRT) is effective for reducing risk of criminal recidivism and improving other health-related outcomes (substance use, mental health, housing, and employment problems) among justice-involved Veterans entering residential mental health treatment programs in the Department of Veterans Affairs (VA).

DETAILED DESCRIPTION:
Approximately 146,000 Veterans are released each year from correctional settings; however, two thirds will likely reoffend and return to the justice system. Antisocial cognitions and behaviors are the strongest predictors of reoffending and are highly prevalent among justice-involved Veterans (JIVs). However, in the absence of treatments with demonstrated effectiveness with JIVs, no systematic approach to address antisocial cognitions and behaviors has been implemented in VA. Moral Reconation Therapy (MRT) is a cognitive-behavioral intervention that aims to reduce antisocial cognitions and behaviors. MRT has the best empirical support for reducing risk for criminal recidivism among civilian offenders, and its associated mechanisms (improvements in interpersonal functioning and impulse control) have been linked to improvements in health-related outcomes that are also risk factors for recidivism (substance use, mental health, housing, and employment problems). However, no trials have been conducted with JIVs. Differences between JIVs and justice-involved civilians (e.g., prevalence of traumatic brain injuries; interpersonal problems) suggests prior research on MRT with civilians may not be generalizable, and prompted the VA's Veterans Justice Programs (VJP) and the developers of MRT to develop a Veteran-specific curriculum of this intervention.

Using the new Veteran-specific manual, the overarching objective of the current proposal is to implement and evaluate MRT as an intervention to reduce risk for criminal recidivism and improve health-related outcomes among JIVs in VA Mental Health Residential Rehabilitation Treatment Programs (MH RRTPs). Using a Hybrid Type 1 design, this project will test the effectiveness of MRT in a multisite Randomized Controlled Trial (RCT) (Palo Alto, Little Rock, and Bedford VAs) and conduct a formative evaluation to facilitate future implementation of MRT in VA.

ELIGIBILITY:
Inclusion Criteria:

* Veterans who

  * (a) are entering a mental health residential rehabilitation treatment program (MH RRTP) at one of three study sites (Palo Alto, Little Rock, or Bedford VA), and
  * (b) had been arrested and charged and/or released from incarceration in the past 5 years prior to MH RRTP admission will be eligible for participation

Exclusion Criteria:

* The only exclusion criterion is being too cognitively impaired to understand the informed consent process and other study procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M. Blonigen, PhD MA, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (3):
- United States (3):
  - Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, North Little Rock, Arkansas
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Timko C, Booth BM, Han X, Schultz NR, Blonigen DM, Wong JJ, Cucciare MA. Criminogenic Needs, Substance Use, and Offending among Rural Stimulant Users. Rural Ment Health. 2017 Apr;41(2):110-122. doi: 10.1037/rmh0000065. PMID 29051795
- [Result] Blonigen DM, Cucciare MA, Timko C, Smith JS, Harnish A, Kemp L, Rosenthal J, Smelson D. Study protocol: a hybrid effectiveness-implementation trial of Moral Reconation Therapy in the US Veterans Health Administration. BMC Health Serv Res. 2018 Mar 7;18(1):164. doi: 10.1186/s12913-018-2967-3. PMID 29514649
- [Result] Blonigen DM, Smith JS, Javier S, Cucciare MA, Timko C, Nevedal AL, Filice N, Rosenthal J, Smelson D. Implementation Potential of Moral Reconation Therapy for Criminal Recidivism in Mental Health Residential Programs. Psychiatr Serv. 2022 Aug 1;73(8):856-863. doi: 10.1176/appi.ps.202100089. Epub 2022 Jan 26. PMID 35080418
- [Result] Blonigen DM, Cucciare MA, Byrne T, Shaffer PM, Giordano B, Smith JS, Timko C, Rosenthal J, Smelson D. A randomized controlled trial of moral reconation therapy to reduce risk for criminal recidivism among justice-involved adults in mental health residential treatment. J Consult Clin Psychol. 2022 May;90(5):413-426. doi: 10.1037/ccp0000721. Epub 2022 Apr 11. PMID 35404638
- [Derived] Ward M, Baldwin N, Blonigen DM. Assessing the impact of combat trauma on the severity, expression, and course of posttraumatic stress disorder in justice-involved veterans. Psychol Trauma. 2025 Jun 2:10.1037/tra0001950. doi: 10.1037/tra0001950. Online ahead of print. PMID 40455528
- [Derived] Timko C, Vest N, Cucciare MA, Smelson D, Blonigen D. Substance use and criminogenic thinking: Longitudinal latent class analysis of veterans with criminal histories. J Subst Abuse Treat. 2022 Dec;143:108893. doi: 10.1016/j.jsat.2022.108893. Epub 2022 Oct 1. PMID 36215912
- [Derived] Gibbon S, Khalifa NR, Cheung NH, Vollm BA, McCarthy L. Psychological interventions for antisocial personality disorder. Cochrane Database Syst Rev. 2020 Sep 3;9(9):CD007668. doi: 10.1002/14651858.CD007668.pub3. PMID 32880104

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on April 4, 2016 from 3 VA Mental Health Residential Rehabilitation Treatment Program (MH RRTP) at Bedford, MA, Little Rock, AR, and Palo Alto, CA. Recruitment officially closed on July 31, 2018.
Pre-assignment Details: A total of 344 participants were enrolled across the 3 sites but only 341 were randomized to either the intervention group or control group. Three participants decided to withdraw from the study for various reasons such as declining to finish the baseline interview or deciding that he/she did not want to participate.
Period: 6-month Follow-up
Arm/Group | Moral Reconation Therapy (MRT) | Usual Care (UC)
Started | 172 | 169
Completed | 119 | 124
Not Completed | 53 | 45
Not completed — Lost to Follow-up | 53 | 45
Period: 12-month Follow-up Interview
Arm/Group | Moral Reconation Therapy (MRT) | Usual Care (UC)
Started | 172 | 169
Completed | 127 | 128
Not Completed | 45 | 41
Not completed — Lost to Follow-up | 45 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moral Reconation Therapy (MRT) | Usual Care (UC) | Total
Number analyzed (Participants) | 172 | 169 | 341
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 166 | 163 | 329
  >=65 years | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.83 (12.191) | 46.60 (12.169) | 46.21 (12.168)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 164 | 161 | 325
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 97 | 100 | 197
  Black or African American | 45 | 52 | 97
  American Indian/Alaska Native | 4 | 2 | 6
  Asian/Pacific Islander | 4 | 2 | 6
  Hispanic or Latino/a, White | 10 | 6 | 16
  Other | 12 | 7 | 19
Controlled environment [Count of Participants; unit: Participants]
  No | 14 | 10 | 24
  Jail | 17 | 10 | 27
  Alcohol or drug treatment | 130 | 135 | 265
  Medical treatment | 2 | 6 | 8
  Psychiatric treatment | 6 | 6 | 12
  Other | 3 | 2 | 5
Sites (U.S.) [Count of Participants; unit: Participants]
  Pacific | 56 | 55 | 111
  Continental | 55 | 55 | 110
  Northeast | 61 | 59 | 120
Days in the residential program [Median (Standard Deviation); unit: Days] | 91.20 (96.035) | 92.55 (100.326) | 91.868 (98.183)

OUTCOME MEASURES:

1. Primary Outcome: Risk for Criminal Recidivism (Criminal Thinking)
Description: The Psychological Inventory of Criminal Thinking Styles (56 items) was administered to assess criminal thinking. The measure includes scales of Mollification, Cutoff, Entitlement, Power Orientation, Super-optimism, Cognitive Indolence, and Discontinuity . Scores on these scales were summed to create a General Criminal Thinking score, which has been validated as an overall index of recidivism risk. Higher scores equate to more criminal thinking. Scores were converted to a T-score metric (M=50, SD=10), calculated in reference to norms from samples of incarcerated offenders.
Time Frame: 6 months (post-baseline)
Population: Intent to treat population (all participants assigned to MRT or UC) analyzed using mixed-effects models. Effectiveness was measured by the time x condition interaction term (UC as the reference group).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Moral Reconation Therapy (MRT) | Usual Care (UC)
Number analyzed (Participants) | 172 | 169
score on a scale | 53.66 [49.2 to 58.1] | 53.30 [48.7 to 58.0]
Statistical Analysis 1: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Models adjusted for covariates (yielded estimated mean values of the outcome) and non-response weights based on completion of follow-up interviews; Time x Condition at 6 mo.(Beta value) = -0.10
Statistical Analysis 2: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); Per protocol analysis, which included all UC participants (n=169) and only those in the MRT condition who had received the minimum recommended dose of the intervention - i.e., Step 3 or higher of MRT (n=63); Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Time x Condition at 6 mo.(Beta value) = -0.88

2. Secondary Outcome: Alcohol Use
Description: The quantity and frequency of patients' self-reported alcohol use in the past 6 months, measured with the Timeline Follow-Back interview that was administered at the 6-month follow-up interview.
Time Frame: 6 months (post-baseline)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of days abstinent (past 6 mo)
Arm/Group | Moral Reconation Therapy (MRT) | Usual Care (UC)
Number analyzed (Participants) | 172 | 169
percentage of days abstinent (past 6 mo) | 94 [90 to 100] | 95 [90 to 100]
Statistical Analysis 1: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Time x Condition at 6 mo.(Beta value) = 0.06
Statistical Analysis 2: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Time x Condition at 6 mo.(Beta value) = 0.02

3. Secondary Outcome: Drug Use
Description: The quantity and frequency of patients' self-reported drug use in the past 6 months, measured with the Timeline Follow-Back interview. It was administered at each time point to calculate for the past 6 months total number of days using any drugs (marijuana, cocaine, amphetamines, heroin, other opiates, benzodiazepines, barbiturates, inhalants, or hallucinogens).
Time Frame: 6 months (post-baseline)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Days (in past 6 months)
Arm/Group | Moral Reconation Therapy (MRT) | Usual Care (UC)
Number analyzed (Participants) | 172 | 169
Days (in past 6 months) | 23.07 [5.0 to 41.1] | 15.01 [-3.7 to 33.7]
Statistical Analysis 1: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Time x Condition at 6 mo.(Beta value) = 10.98
Statistical Analysis 2: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Time x Condition at 6 mo.(Beta value) = 14.64

4. Secondary Outcome: Criminal Associates
Description: Scale A of the Measures of Criminal Attitudes and Associates (MCAA; Mills, Kroner, & Forth, 2002) was administered at each interview to quantify participants' associations with criminal peers, a strong predictor of criminal recidivism (Mills, Kroner, & Hemmati, 2004). Participants were asked to consider the four adults (excluding family, co-workers, or other residents in treatment) with whom they spend the most free-time. A count variable was created by summing the number of friends for which the participant answered yes to any of the questions of criminal involvement (possible range=0-4, where a higher score indicates a worse outcome)
Time Frame: 6 months (post-baseline)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: friends with criminal involvement
Arm/Group | Moral Reconation Therapy (MRT) | Usual Care (UC)
Number analyzed (Participants) | 172 | 169
friends with criminal involvement | 0.43 [0.2 to 0.8] | 0.28 [0.1 to 0.6]
Statistical Analysis 1: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Time x Condition at 6 mo.(Beta value) = 1.45
Statistical Analysis 2: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Time x Condition at 6 mo.(Beta value) = 1.22

5. Secondary Outcome: Employment Problem Severity
Description: The Employment module of the ASI was administered at each timepoint to assess problem severity in this domain, using composite score indices (range 0 to 1); higher scores indicate greater problem severity.
Time Frame: 6 months (post-baseline)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Moral Reconation Therapy (MRT) | Usual Care (UC)
Number analyzed (Participants) | 172 | 169
score on a scale | 0.58 [0.5 to 0.7] | 0.61 [0.5 to 0.7]
Statistical Analysis 1: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Time x Condition at 6 mo.(Beta value) = 0.04
Statistical Analysis 2: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Time x Condition at 6 mo.(Beta value) = 0.02

6. Secondary Outcome: Alcohol Use Problem Severity.
Description: The Alcohol module of the ASI was administered at each time point to assess problem severity in this domain, using composite score indices (ranging from 0 to 1); higher scores indicate greater problem severity. ASI composite scores such as this have long been used to provide internally-consistent evaluations of a patient in a particular problem area (Grahn & Padyab, 2020).
Time Frame: 6 months (post-baseline)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Moral Reconation Therapy (MRT) | Usual Care (UC)
Number analyzed (Participants) | 172 | 169
score on a scale | 0.09 [0.0 to 0.2] | 0.06 [0.0 to 0.1]
Statistical Analysis 1: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Time x Condition at 6mo.(Beta value) = 0.04
Statistical Analysis 2: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Time x Condition at 6 mo.(Beta value) = 0.02

7. Secondary Outcome: Legal Problem Severity
Description: The Legal Status module of the Addiction Severity Index (ASI; McLellan et al., 2006) was administered at each interview to assess legal problem severity. The latter is based on a composite index derived from five items: Are you presently awaiting charges, trial, or sentence? How many days in the past 30 have you engaged in illegal activities for profit? How serious do you feel your present legal problems are? (0=Not at all, 4=Extremely) How important to you now is counseling or referral for these legal problems? (0=Not at all, 4=Extremely) How much money did you receive from illegal sources in the past 30 days? These items were standardized and aggregated and yield scores ranging from 0 to 1; higher scores indicate greater problem severity of legal problems.
Time Frame: 6 months (post-baseline)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Moral Reconation Therapy (MRT) | Usual Care (UC)
Number analyzed (Participants) | 172 | 169
score on a scale | 0.14 [0.10 to 0.20] | 0.13 [0.10 to 0.20]
Statistical Analysis 1: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Time x Condition at 6 mo.(Beta value) = 0.02
Statistical Analysis 2: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Time x Condition at 6 mo.(Beta value) = -0.08

8. Secondary Outcome: Family/Social Problems
Description: The Family/Social module of the ASI was administered at each timepoint to assess problem severity in this domain, using composite score indices (range 0 to 1); higher scores indicate greater problem severity.
Time Frame: 6 months (post-baseline)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Moral Reconation Therapy (MRT) | Usual Care (UC)
Number analyzed (Participants) | 172 | 169
score on a scale | 0.1 [0.1 to 0.2] | 0.1 [0.0 to 0.2]
Statistical Analysis 1: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); Test type: Superiority; p < 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Time x Condition at 6 mo.(Beta value) = 0.06
Statistical Analysis 2: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Time x Condition at 6 mo.(Beta value) = 0.06

9. Primary Outcome: Risk for Criminal Recidivism (Criminal Thinking)
Description: as for outcome 1
Time Frame: 12 months (post-baseline)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Moral Reconation Therapy (MRT) | Usual Care (UC)
Number analyzed (Participants) | 172 | 169
score on a scale | 50.96 [46.5 to 55.4] | 49.80 [45.2 to 54.4]
Statistical Analysis 1: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Other[Time x Condition at 12 mo.(Beta = 0.69
Statistical Analysis 2: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Other[Time x Condition at 12 mo.(Beta v = -0.89

10. Secondary Outcome: Alcohol Use
Description: The quantity and frequency of patients' self-reported alcohol use in the past 6 months, measured with the Timeline Follow-Back interview that was administered at the 12-month follow-up interview.
Time Frame: 12 months (post-baseline)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of days abstinent (past 6 mo)
Arm/Group | Moral Reconation Therapy (MRT) | Usual Care (UC)
Number analyzed (Participants) | 172 | 169
percentage of days abstinent (past 6 mo) | 94 [90 to 100] | 94 [90 to 100]
Statistical Analysis 1: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Other[Time x Condition at 12 mo.(Beta v = 0.07
Statistical Analysis 2: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Other[Time x Condition at 12 mo.(Beta v = 0.01

11. Secondary Outcome: Drug Use
Description: as for outcome 3
Time Frame: 12 months (post-baseline)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Days (in past 6 months)
Arm/Group | Moral Reconation Therapy (MRT) | Usual Care (UC)
Number analyzed (Participants) | 172 | 169
Days (in past 6 months) | 18.63 [0.4 to 36.8] | 15.03 [-3.6 to 33.6]
Statistical Analysis 1: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Other[Time x Condition at 12 mo.(Beta v = 6.53
Statistical Analysis 2: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); Per protocol analysis, which included all UC participants (n=169) and only those in the MRT condition who had received the minimum recommended dose of the intervention - i.e., Step 3 or higher of MRT (n=63; Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Other[Time x Condition at 12 mo.(Beta v = 5.68

12. Secondary Outcome: Criminal Associates
Description: as for outcome 4
Time Frame: 12 months (post-baseline)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: friends with criminal involvement
Arm/Group | Moral Reconation Therapy (MRT) | Usual Care (UC)
Number analyzed (Participants) | 172 | 169
friends with criminal involvement | 0.37 [0.2 to 0.7] | 0.43 [0.2 to 0.8]
Statistical Analysis 1: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Other[Time x Condition at 12 mo.(Beta v = 0.83
Statistical Analysis 2: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.01, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Other[Time x Condition at 12 mo.(Beta v = 0.46

13. Secondary Outcome: Employment Problem Severity
Description: as for outcome 5
Time Frame: 12 months (post-baseline)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Moral Reconation Therapy (MRT) | Usual Care (UC)
Number analyzed (Participants) | 172 | 169
score on a scale | 0.48 [0.4 to 0.6] | 0.53 [0.4 to 0.6]
Statistical Analysis 1: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Other[Time x Condition at 12 mo.(Beta) = 0.02
Statistical Analysis 2: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Other[Time x Condition at 12 mo.(Beta) = -0.08

14. Secondary Outcome: Alcohol Use Problem Severity.
Description: as for outcome 6
Time Frame: 12 months (post-baseline)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Moral Reconation Therapy (MRT) | Usual Care (UC)
Number analyzed (Participants) | 172 | 169
score on a scale | 0.04 [0.0 to 0.1] | 0.06 [0.0 to 0.1]
Statistical Analysis 1: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Other[Time x Condition at 12 mo.(Beta)] = -0.03
Statistical Analysis 2: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Other[Time x Condition at 12 mo.(Beta)] = -0.07

15. Secondary Outcome: Legal Problem Severity
Description: as for outcome 7
Time Frame: 12 months (post-baseline)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Moral Reconation Therapy (MRT) | Usual Care (UC)
Number analyzed (Participants) | 172 | 169
score on a scale | 0.09 [0.03 to 0.15] | 0.09 [0.02 to 0.15]
Statistical Analysis 1: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Other[Time x Condition at 12 mo.(Beta)] = 0.01
Statistical Analysis 2: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Other[Time x Condition at 12 mo.(Beta)] = -0.08

16. Secondary Outcome: Family/Social Problems
Description: as for outcome 8
Time Frame: 12 months (post-baseline)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Moral Reconation Therapy (MRT) | Usual Care (UC)
Number analyzed (Participants) | 172 | 169
score on a scale | 0.19 [0.1 to 0.2] | 0.11 [0.1 to 0.2]
Statistical Analysis 1: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); Test type: Superiority; p < 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Other[Time x Condition at 12 mo.(Beta)] = 0.07
Statistical Analysis 2: Comparison: Moral Reconation Therapy (MRT) vs Usual Care (UC); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Other[Time x Condition at 12 mo.(Beta)] = 0.08

ADVERSE EVENTS:
Time Frame: Adverse event data was collected in the 12 months post-baseline for each participant.
Arm/Group | Moral Reconation Therapy (MRT) | Usual Care (UC)
All-Cause Mortality (participants affected / at risk) | 7/172 | 12/169
Serious Adverse Events (participants affected / at risk) | 2/172 | 4/169
Other Adverse Events (participants affected / at risk) | 0/172 | 0/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moral Reconation Therapy (MRT) (N=172) | Usual Care (UC) (N=169)
Death (Social circumstances) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT02524171/Prot_SAP_000.pdf
  • Informed Consent Form (2016-09-16): https://cdn.clinicaltrials.gov/large-docs/71/NCT02524171/ICF_001.pdf